CLINICAL TRIAL: NCT00056147
Title: Multi-Center, Double-Blind, Randomized, Placebo-Controlled, 28-Day Study of INS37217 Inhalation Solution in Subjects With Mild to Moderate Cystic Fibrosis Lung Disease
Brief Title: Study of INS37217 Inhalation Solution in Mild to Moderate Cystic Fibrosis Lung Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-103
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — denufosol tetrasodium

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217)

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of multiple dosages of INS37217 compared to placebo over 28 days in subjects with mild to moderate cystic fibrosis (CF) lung disease. Study drug will be administered through a nebulizer (a device that delivers medication as a mist by breathing it in).

DETAILED DESCRIPTION:
The purpose of this study is to:

* assess the safety and efficacy of multiple dose levels of INS37217 compared to placebo over 28 days in subjects with mild to moderate CF lung disease;
* explore evidence of activity of INS37217 and placebo administered via PARI LC STAR nebulizer;
* identify dose(s) that will be studied in subsequent trials.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of CF
* FEV1 greater than or equal to 75% of predicted normal for age, gender, and height
* oxyhemoglobin saturation greater than or equal to 90%
* clinically stable

Exclusion Criteria:

* abnormal renal or liver function
* clinically significant findings atypical for moderate cystic fibrosis

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2003-04; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
lung function
respiratory symptoms
sputum weight
pulmonary exacerbations
measures of lung characteristics

SECONDARY OUTCOMES:
safety measures

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director

REFERENCES:
- [Result] Deterding RR, Lavange LM, Engels JM, Mathews DW, Coquillette SJ, Brody AS, Millard SP, Ramsey BW; Cystic Fibrosis Therapeutics Development Network and the Inspire 08-103 Working Group. Phase 2 randomized safety and efficacy trial of nebulized denufosol tetrasodium in cystic fibrosis. Am J Respir Crit Care Med. 2007 Aug 15;176(4):362-9. doi: 10.1164/rccm.200608-1238OC. Epub 2007 Apr 19. PMID 17446337